CLINICAL TRIAL: NCT03223012
Title: Post-marketing Prospective, Observational Cohort Study to Evaluate the Impact of AbbVie Care Patient Support Program on Compliance With Adalimumab, Patient Reported Outcomes and Health Resource Utilization in Inflammatory Bowel Diseases, Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis and Psoriasis in Portugal
Brief Title: Impact of AbbVie Care Patient Support Program on Clinical, Health Economic and Patient Reported Outcomes, in Crohn's Disease, Ulcerative Colitis, Rheumatoid Arthritis, Psoriatic Arthritis, Psoriasis and Axial Spondyloarthritis, in the Portuguese National Health Service
Acronym: IMPROVE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-321
Record Dates: First submitted 2017-07-18; First posted 2017-07-19 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Crohn's Disease; Ulcerative Colitis (UC); Rheumatoid Arthritis (RA); Psoriatic Arthritis; Psoriasis; Ankylosing Spondylitis (AS); Non-radiographic Axial Spondyloarthritis
Keywords: Adalimumab; Humira®; AbbVie patient care support program; Psoriasis; Axial Spondyloarthritis; Rheumatoid Arthritis; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Arthritis, Rheumatoid; Arthritis, Psoriatic; Psoriasis; Spondylitis, Ankylosing; Non-Radiographic Axial Spondyloarthritis; Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants not included in the AbbVie care program: Participants receiving adalimumab not included in the AbbVie care patient support program.
- Participants included in the AbbVie care program: Participants receiving adalimumab included in the AbbVie care patient support program.

SUMMARY:
This study aims to evaluate the impact of AbbVie Care 2.0 on adalimumab's compliance, patient reported outcomes and utilization of health resources over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with crohn's disease (CD), ulcerative colitis (UC), rheumatoid arthritis (RA), psoriatic arthritis (PsA), axial spondyloarthritis (SpA) or psoriasis (Pso) according to the treating physician
* Adalimumab was started within 1 month prior to study enrollment
* Adalimumab was introduced based on current clinical practice criteria (i.e., the prescription of adalimumab was clearly separated from the decision to include the participants in this study)
* No prior record of adalimumab treatment
* Adalimumab was administered according to product label
* Naïve or previously experienced with biologic treatment
* Participant is able and willing to provide written authorization to disclose and use personal health information (informed consent), and to agree that data will be collected and provided to AbbVie

AbbVie Care 2.0 Cohort-specific inclusion criteria:

* Initiated the AbbVie care program within the first month after starting adalimumab.

Exclusion Criteria:

* Definitive discontinuation of adalimumab before being proposed to participate in the study
* Participated in any clinical experimental research within the 2 months prior to enrollment
* Pregnant or breastfeeding female participants
* Participant not able or not willing to comply with the requirements of this study protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants receiving adalimumab in routine clinical practice in Portugal
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Medication Possession Ratio (MPR)>=80% | Up to 12 months
  The variable MPR will be used, considering in the numerator the sum of days supply between start of observation (baseline) and last prescription dispensed (including the days of last prescription) and as denominator the number of days elapsed between baseline and last prescription dispensed (including the days of last prescription).

SECONDARY OUTCOMES:
Mean number of injections administered/ prescribed for adalimumab | Up to 12 months
  This is assessed based on patient diary.
Assessing Patient's overall satisfaction with AbbVie Care 2.0 program | At 12 months
  Patient's overall satisfaction with AbbVie Care 2.0 program is scored at 1: Very good, 2: Good and 3: Less satisfying.
Number of Sick Leaves | Up to 12 months
  This is assessed by reviewing work time lost due to other reasons than health problems during previous last seven days.
Time Spent by the Patient to Refill Prescription | Up to 12 months
  This is assessed by reviewing the work productivity indicator over 12 months.
Number of Hospital Inpatient Days | Up to 12 months
  This is assessed by reviewing the use of health resources over 12 months.
Number of Emergency Visits | Up to 12 months
  This is assessed by reviewing the use of health resources over 12 months.
Assessing Working Status | Up to 12 months
  This is assessed by the proportion of patients employed.
Proportion of patients with MPR>=80% | At Month 6
  The variable MPR will be used, considering in the numerator the sum of days supply between start of observation (baseline) and last prescription dispensed (including the days of last prescription) and as denominator the number of days elapsed between baseline and last prescription dispensed (including the days of last prescription).
Mean score of Treatment Satisfaction Questionnaire for Medication (TSQM)-II | Up to Month 12
  This 14-point measure attempts to show that adherence is expected to be related with patients' satisfaction with therapy and such satisfaction can be a function of not only the effect of the treatment, but also the services offered. Domains include: Effectiveness, Side effects, Convenience and Global satisfaction.
Mean Change in EuroQoL (EQ-5D) score | From Month 0 to Month 12
  EQ-5D considers five attributes of quality of life evaluation, i.e., mobility, self-care, usual activity, pain/ discomfort, and anxiety/ depression.
Number of Complementary Exams/ Techniques | Up to 12 months
  This is assessed by reviewing the use of health resources over 12 months.
Number of Hospitalizations | Up to 12 months
  This is assessed by reviewing the use of health resources over 12 months.
Time Spent by the Health Care Providers (HCPs) During Medical Appointments | Up to 12 months
  This is assessed by reviewing the use of health resources over 12 months.
Mean Change in Patient Activation Measure (PAM-13) | From Month 0 to Month 12
  This is a powerful and reliable measure of patient activation. It is 13-item measure used to assess the patient knowledge, skill, and confidence for self-management.
Mean Change in Beliefs about Medication Questionnaire (BMQ) | From Month 0 to Month 12
  The BMQ comprises two sections: the BMQ-Specific, which assesses representations of medication prescribed for personal use and the BMQ-General, which assesses beliefs about medicines in general. This questionnaire is validated for use in Portugal.
Change in Work Productivity and Activity Impairment- General Health (WPAI-GH) | From Month 0 to Month 12
  WPA-GH assesses the impact of general health problem on work productivity and daily activities during the previous 7 days.
Number of Outpatient Visits (in-office and remote) in Hospital Setting | Up to 12 months
  This is assessed by reviewing the use of health resources over 12 months.
Number of Days of Sick Leaves | Up to 12 months
  This is assessed by reviewing work time lost due to health problems during previous seven days.
Proportion of patients who are still on adalimumab after 6 and 12 months | Up to 12 months
  This is used to assess persistence and it could be done using pharmacy refills.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (15):
- Portugal (15):
  - Instituto Portugues De Reumatologia /ID# 205963, Lisbon, Lisbon District
  - Centro Hosp de Lisboa Central /ID# 205698, Lisbon, Lisbon District
  - Centro Hospitalar Lisboa Ocidental, EPE /ID# 201328, Lisbon, Lisbon District
  - Centro Hospitalar Lisboa Ocidental, EPE /ID# 201330, Lisbon, Lisbon District
  - CCA Braga - Hospital de Braga /ID# 201322, Braga
  - CCA Braga - Hospital de Braga /ID# 201323, Braga
  - CCA Braga - Hospital de Braga /ID# 201324, Braga
  - Hospital Santo Antonio dos Cap /ID# 205700, Lisbon
  - Centro Hospitalar Lisboa Norte, EPE /ID# 201335, Lisbon
  - Centro Hospitalar Lisboa Norte, EPE /ID# 201336, Lisbon
  - Centro Hospitalar Lisboa Norte, EPE /ID# 201337, Lisbon
  - Centro Hospitalar de Sao Joao, EPE /ID# 203535, Porto
  - Centro Hospitalar de Sao Joao, EPE /ID# 206278, Porto
  - Centro Hosp de Tondela-Viseu /ID# 203774, Viseu
  - Centro Hosp de Tondela-Viseu /ID# 203775, Viseu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P16-321.pdf